CLINICAL TRIAL: NCT01783873
Title: Comparative Study of Pathophysiological Mechanisms and Bronchial Response in Occupational Asthma to Wheat Flour and Quaternary Ammonium Compounds During Standardized Bronchial Provocation Tests
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitement difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 4707
Record Dates: First submitted 2013-01-28; First posted 2013-02-05 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2019-08

CONDITIONS: Occupational Asthma
MeSH Terms: conditions — Asthma, Occupational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: standardized bronchial challenge test (SCL SCL • • GenaSOL ™ GenaSIC ™)
- flour allergen extract or quaternary ammonium compound (Active Comparator)
  Interventions: Other: standardized bronchial challenge test (SCL SCL • • GenaSOL ™ GenaSIC ™)

INTERVENTIONS:
Other: standardized bronchial challenge test (SCL SCL • • GenaSOL ™ GenaSIC ™) — At Visit 1: Patients are selected and they will receive a metacholine challenge test during and outside of work. After randomization, patients undergo a standardized bronchial challenge test (SCL SCL • • GenaSOL ™ GenaSIC ™) to either an wheat flour allergen extract or didecyldimethylammonium chloride or placebo. Each bronchial challenge test is followed by blood sampling at different time points and induced sputum. The immediate bronchial response and late bronchial response will be recorded.

SUMMARY:
Occupational asthma (OA) caused by high molecular weight (HMW) substances have been shown to induce predominantly an eosinophilic inflammation. In contrast, OA caused by low molecular weight (LMW) substances results in a neutrophilic inflammation. In addition, data regarding phenotype of lymphocytes in OA caused by HMW and LMW substances are scarce. The use of a new equipment will allow the realization of specific standardized bronchial challenges (BC) to occupational agents. Thus, we propose to study in more detail the cellular mechanisms involved during BC to HMW and LMW occupational agents in a double-blind placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

For patients with occupational asthma to wheat flour:

* Clinical history,
* A positive skin test to wheat flour and / or specific IgE to wheat flour

For patients with occupational asthma to quaternary ammonium compounds:

-Clinical history,

For two types of asthma:

* Patients must have a worsening of bronchial hyperreactivity during work compared to a rest period assessed by a metacholine challenge
* FEV before challenge (nonspecific and specific) must be> 70%.

Exclusion Criteria:

Asthmas:

* no occupational asthma:
* secondary to clinically relevant sensitization to an allergen domestic
* aggravated at work.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09; Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Assessment of cellular inflammation in peripheral blood and induced sputum | 33 months
  Before and after bronchial challenge: assessment of cellular inflammation in peripheral blood and induced sputum, exhaled NO; assessment of peripheral T lymphocyte phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric De BLAY, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France